CLINICAL TRIAL: NCT00514943
Title: A Randomized, Open-label Phase II Study of BIBW 2992 Versus Cetuximab (Erbitux) in Patients With Metastatic or Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC) After Failure of Platinum-containing Therapy With a Cross-over Period for Progressing Patients
Brief Title: BIBW 2992 (Afatinib) in Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1200.28; 2008-007097-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Afatinib; Cetuximab

ARMS (2):
- BIBW 2992 (Experimental): once daily taken orally
  Interventions: Drug: BIBW 2992
- Cetuximab (Active Comparator): once every week by intravenous injection
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: BIBW 2992 — experimental drug taken once daily orally
  Arms: BIBW 2992
Drug: Cetuximab — active comparator administered weekly intravenously
  Arms: Cetuximab

SUMMARY:
The primary objective of this study is to explore the efficacy of BIBW 2992 compared with cetuximab (Erbitux) in patients with metastatic or recurrent head and neck cancer after failure of platinum-containing therapy. In addition, the trial aims to clarify the influence of EGFR genotype on tumor response to the treatment regimens.

ELIGIBILITY:
Inclusion criteria:

1. Metastatic (stage IVc) or recurrent HNSCC 2. Histologically or cytologically confirmed diagnosis of squamous cell of the head and neck. Patients with well-differentiated (keratinizing) nasopharyngeal carcinomas and patients with squamous cell carcinomas metastatic to the neck from an unknown head and neck primary are eligible. 3. Patients must have documented progressive disease (PD) following receipt of prior platinum-based therapy (either as neoadjuvant, adjuvant, concomitant with radiotherapy, or for recurrent/ metastatic disease). 4. Patients must have measurable disease as defined by RECIST criteria. 5. Patients must have recovered from any therapy-related toxicities from previous chemo-, immuno-, or radiotherapies to CTC smaller or equal to Grade 1. 6. Patients must have recovered from previous surgery. 7. Life expectancy of at least three (3) months. 8. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score 0 or 1.

9. Patients must be eighteen (18) years of age or older. 10. Willingness and ability to give written informed consent consistent with ICH-GCP guidelines.

Exclusion criteria:

1. Progressive disease within 3 months after completion of curative intent treatment for localized/locoregionally advanced disease.
2. Prior use of an EGFR or erbB2 inhibitor in the recurrent/metastatic disease setting (treatment with cetuximab (Erbitux®) or other EGFR inhibitor during radiotherapy or chemoradiotherapy is permissible).
3. More than 2 chemotherapeutic regimens given for recurrent/metastatic disease.
4. Treatment with other investigational drugs, other anti-cancer-therapy (e.g., chemotherapy, immunotherapy, radiotherapy), concomitantly with therapy on this study and/or during the last four weeks, prior to the first treatment with the trial drug
5. eliminated per Amendment #1
6. Patients with history of other malignancy (except for appropriately treated superficial basal cell skin cancer and surgically cured cervical cancer in situ) unless free of disease for at least 3 years.
7. Patients with history of decompensated heart failure.
8. Cardiac left ventricular function with resting ejection fraction <50% or less than the institutional lower limit of normal by MUGA or echocardiogram.
9. Active infectious disease.
10. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea.
11. Serious illness, concomitant non-oncological disease or mental problems considered by the investigator to be incompatible with the protocol.
12. Use of alcohol or drugs incompatible with patient participation in the study in the investigator's opinion.
13. Patients unable to comply with the protocol.
14. Patients with active/symptomatic brain metastases. Patients with a history of treated brain metastases must have stable or normal cerebral MRI scan at screening and be at least three months post-radiation or surgery.
15. Absolute neutrophile count (ANC) less than 1000/mm3.
16. Platelet count less than 75,000/mm3.
17. Bilirubin greater than 1.5 mg/dl/ Higher bilirubin values are acceptable for patients with known Gilbert's disease, approval by the PI and sponsor necessary.
18. Asparate amino transferase (AST) or alanine amino transferase (ALT) greater than 3 times the upper limit of normal.
19. Serum creatinine greater than 1.5 X upper limit of normal for the institution.
20. Patients who are sexually active and unwilling to use a medically acceptable method of contraception.
21. Pregnancy or breast-feeding.
22. Patients with known pre-existing interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- United States (18):
  - 1200.28.0010 Boehringer Ingelheim Investigational Site, Stanford, California
  - 1200.28.0001 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1200.28.0005 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1200.28.0011 Boehringer Ingelheim Investigational Site, Harvey, Illinois
  - 1200.28.0022 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1200.28.0024 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1200.28.0012 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1200.28.0021 Boehringer Ingelheim Investigational Site, Saint Joseph, Michigan
  - 1200.28.0016 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 1200.28.0002 Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - 1200.28.0006 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1200.28.0008 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1200.28.0017 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1200.28.0004 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1200.28.0013 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1200.28.0007 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1200.28.0009 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1200.28.0020 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Belgium (3):
  - 1200.28.0030 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.28.0031 Boehringer Ingelheim Investigational Site, Ghent
  - 1200.28.0032 Boehringer Ingelheim Investigational Site, Leuven
- France (9):
  - 1200.28.0062A Boehringer Ingelheim Investigational Site, Alès
  - 1200.28.0062B Boehringer Ingelheim Investigational Site, Alès
  - 1200.28.0059A Boehringer Ingelheim Investigational Site, Avignon
  - 1200.28.0052A Boehringer Ingelheim Investigational Site, Lille
  - 1200.28.0051A Boehringer Ingelheim Investigational Site, Lyon
  - 1200.28.0050A Boehringer Ingelheim Investigational Site, Montpellier
  - 1200.28.0058A Boehringer Ingelheim Investigational Site, Nîmes
  - 1200.28.0061A Boehringer Ingelheim Investigational Site, Poitiers
  - 1200.28.0055G Boehringer Ingelheim Investigational Site, Rouen
- Spain (6):
  - 1200.28.0040 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.28.0044 Boehringer Ingelheim Investigational Site, Barcelona
  - 1200.28.0043 Boehringer Ingelheim Investigational Site, Madrid
  - 1200.28.0042 Boehringer Ingelheim Investigational Site, Málaga
  - 1200.28.0045 Boehringer Ingelheim Investigational Site, Santander
  - 1200.28.0041 Boehringer Ingelheim Investigational Site, Valencia

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label randomized, cross-over study. 124 patients were randomised. 3 patients were not treated, 1 in Afatinib arm and 2 in Cetuximab arm.
Groups:
- Afatinib 50 mg / Cetuximab 250mg/m2: Patients were randomized to Afatinib monotherapy 50mg once daily (q.d.) in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week (load) followed by 250mg/m2 weekly thereafter in Stage 2.
- Cetuximab 250 mg/m2 / Afatinib 50 mg: Patients were randomized to Cetuximab 250 mg/m2 received 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Afatinib 50 mg once daily (q.d.) for Stage 2
Period: Stage 1
Arm/Group | Afatinib 50 mg / Cetuximab 250mg/m2 | Cetuximab 250 mg/m2 / Afatinib 50 mg
Started | 62 (1 randomized patient was not treated) | 62 (2 randomized patients were not treated)
Completed | 32 | 36
Not Completed | 30 | 26
Not completed — Progressive disease | 4 | 8
Not completed — Other Adverse Event | 16 | 6
Not completed — Not treated | 1 | 2
Not completed — Patient refused to continue study meds | 8 | 3
Not completed — Other than stated above | 1 | 7
Period: Stage 2
Arm/Group | Afatinib 50 mg / Cetuximab 250mg/m2 | Cetuximab 250 mg/m2 / Afatinib 50 mg
Started | 32 | 36
Completed | 0 | 0
Not Completed | 32 | 36
Not completed — Progressive disease | 27 | 24
Not completed — Other Adverse Event | 3 | 10
Not completed — Patient refused to continue study meds | 2 | 0
Not completed — Other than stated above | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 50 mg / Cetuximab 250mg/m2 | Cetuximab 250 mg/m2 / Afatinib 50 mg | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.4) | 58.8 (8.7) | 58.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 55 | 52 | 107
Prior chemotherapies (CT)for recurrent/metastatic disease (R/M) [Number; unit: Number of participants]
  Yes | 42 | 41 | 83
  No | 20 | 21 | 41
Baseline sum of longest diameters (SLD) of target lesions by investigator assessments [Mean (Standard Deviation); unit: millimeters] — Baseline measures were available for only 61 patients in the Afatinib/Cetuximab group and only 60 patients in the Cetuximab/Afatinib group
  millimeters | 71.4 (44.6) | 65.4 (44.2) | 68.4 (44.3)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Shrinkage Before Crossover (Stage 1) of the Trial as Per Investigator Assessment
Description: Tumor shrinkage before crossover was defined as the change from baseline in the smallest post-randomisation sum of the longest diameters of target lesions (SLD), calculated as the smallest SLD after randomisation but before crossover minus SLD at baseline. Baseline was the SLD measured before randomisation. A negative value means the smallest post-randomisation SLD was smaller than baseline (decreased since baseline); a positive value means tumor size increased since baseline.
  Mean calculated is actually the Adjusted mean. Adjusted mean is obtained from fitting an ANCOVA model including treatment, stratification factor prior chemotherapy for recurrent/metastatic disease and the baseline sum of longest distance of target lesions as covariates.
Time Frame: From randomization until start of Stage 2 treatment, or within 28 days after the termination of Stage 1.
Population: Randomised Set (RS). The randomised set includes all patients who were randomised to receive treatment, whether treated or not. However, patients without baseline or post-baseline tumor measurements were excluded.
Measure: Mean (Standard Error); unit: millimeter
Groups:
- Afatinib 50 mg - Stage 1: Patients were randomised to receive Afatinib 50 mg once daily (q.d.) in Stage 1.
- Cetuximab 250 mg/m2 - Stage 1: Patients were randomized to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1.
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 50 | 55
millimeter | -3.86 (3.62) | -2.37 (3.47)
Statistical Analysis 1: Comparison: Afatinib 50 mg - Stage 1 vs Cetuximab 250 mg/m2 - Stage 1; Test type: Superiority or Other; p = 0.7606, ANCOVA — P-value obtained from fitting an ANCOVA model including treatment, stratification factor prior chemotherapy for recurrent/metastatic disease and the baseline sum of longest distance of target lesions; Receipt of prior chemotherapy for recurrent/metastatic disease and the baseline sum of longest distance for target lesions are covariates; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-11.188 to 8.202] — Mean difference calculated is actually the adjusted mean difference

2. Secondary Outcome: Tumor Shrinkage After Crossover (Stage 2) as Per Investigator Assessments
Description: Tumor shrinkage after crossover was defined as the change from baseline in the smallest post-crossover sum of the longest diameters of target lesions (SLD), calculated as the smallest SLD after crossover minus SLD at baseline. Baseline was the SLD measured at the time of crossover, or the closest measurement before the patient started stage 2 treatment. A negative value means the smallest post-crossover SLD was smaller than baseline (decreased after crossover), a positive value means tumor size increased after crossover.
Time Frame: From baseline assessed prior to first dose of Stage 2 study medication to 28 days after termination of Stage 2 treatment.
Population: Patients treated in stage 2 : This analysis set included all patients who received treatment: 36 patients in the afatinib and 32 patients in the cetuximab arm.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Afatinib 50 mg - Stage 2: Patients were randomized to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Afatinib 50 mg once daily (q.d.) for Stage 2
- Cetuximab 250 mg/m2 - Stage 2: Patients were randomized to Afatinib monotherapy 50mg once daily (q.d.) in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week (load) followed by 250mg/m2 weekly thereafter in Stage 2.
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 29 | 27
millimeters | 2 (15) | 16 (30)

3. Secondary Outcome: Best RECIST Assessment as Per Investigator Assessment for Stage 1 (as Confirmed Disease Control (Clinical Benefit) and Objective Response Are Simply Categories of RECIST Assessment).
Description: Best RECIST Assessment is defined as confirmed Disease control (complete response (CR), partial response (PR) and Stable disease (SD)), Objective response ( complete response (CR) or partial response (PR)) assessed by the investigator according to the RECIST 1.0 criteria.
Time Frame: Response determined from randomization until patient started Stage 2 or within 28 days after termination of Stage 1 treatment
Population: Randomised set (RS).
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
Number of participants
  Disease control (CR, PR, SD) | 31 | 35
  Objective response (CR, PR) | 10 | 4
  Complete response (CR) | 0 | 2
  Partial response (PR) | 10 | 2
  Stable disease (SD) | 21 | 31
  Progressive disease (PD) | 16 | 19
  Not evaluable | 5 | 1
  Missing | 10 | 7

4. Secondary Outcome: Best RECIST Assessment as Per ICR for Stage 1 (as Confirmed Disease Control (Clinical Benefit) and Objective Response Are Simply Categories of RECIST Assessment).
Description: Best RECIST Assessment is defined as confirmed Disease control (complete response (CR), partial response (PR) and Stable disease (SD)), Best objective response ( complete response (CR) or partial response (PR)) as assessed by the independent central review (ICR) according to the RECIST 1.0 criteria.
Time Frame: as for outcome 3
Population: Randomised set (RS).
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
Number of participants
  Disease control (CR, PR, SD) | 29 | 30
  Objective response (CR,PR) | 5 | 6
  Complete response (CR) | 0 | 0
  Partial response (PR) | 5 | 6
  Stable disease (SD) | 24 | 24
  Progressive disease (PD) | 21 | 21
  Not evaluable | 2 | 3
  Missing | 10 | 8

5. Secondary Outcome: Best RECIST Assessment as Per Investigator Assessment for Stage 2 (as as Confirmed Disease Control (Clinical Benefit) and Objective Response Are Simply Categories of RECIST Assessment)
Description: as for outcome 3
Time Frame: Response determined during Stage 2 or within 28 days after termination of Stage 2 treatment
Population: Patients treated in Stage 2
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 36 | 32
Number of participants
  Disease control (CR, PR, SD) | 14 | 6
  Objective response (CR,PR) | 1 | 2
  Complete response (CR) | 1 | 0
  Partial response (PR) | 0 | 2
  Stable disease (SD) | 13 | 4
  Progressive disease (PD) | 16 | 20
  Not evaluable | 1 | 4
  Missing | 5 | 2

6. Secondary Outcome: Best RECIST Assessment as Per ICR for Stage2 (as Confirmed Disease Control (Clinical Benefit) and Objective Response Are Simply Categories of RECIST Assessment)
Description: as for outcome 4
Time Frame: Response determined during Stage 2 or within 28 days after termination of Stage 2 treatment
Population: Patients treated in Stage 2
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 36 | 32
Number of participants
  Disease control (CR, PR, SD) | 12 | 6
  Objective response | 0 | 0
  Complete response (CR) | 0 | 0
  Partial response (PR) | 0 | 0
  Stable disease (SD) | 12 | 6
  Progressive disease (PD) | 18 | 21
  Not evaluable | 1 | 4
  Missing | 5 | 1

7. Secondary Outcome: Best RECIST Assessment as Onset of Confirmed Objective Response as Per Investigator Assessment for Stage 1
Description: Best RECIST Assessment as onset of confirmed objective response as per Investigator assessment for Stage 1.
Time Frame: as for outcome 3
Population: Randomised set (RS).
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 10 | 4
Number of participants
  Week 4 (Day 1 - 42) | 3 | 0
  Week 8 (Day 43 - 84) | 1 | 3
  Week 16 (Day 85 - 140) | 4 | 1
  Week 24 (Day 141 - 196) | 2 | 0

8. Secondary Outcome: Best RECIST Assessment as Onset of Confirmed Objective Response as as Per ICR for Stage 1
Description: Best RECIST Assessment as onset of confirmed objective response as per the independent central review (ICR) according to the RECIST 1.0 criteria.
Time Frame: as for outcome 3
Population: Randomised set (RS).
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 5 | 6
Number of participants
  Week 4 (Day 1 - 42) | 1 | 0
  Week 8 (Day 43 - 84) | 2 | 3
  Week 16 (Day 85 - 140) | 2 | 2
  Week 24 (Day 141 - 196) | 0 | 1

9. Secondary Outcome: Best RECIST Assessment as Onset of Confirmed Objective Response as Per Investigator Assessment for Stage 2
Description: Best RECIST Assessment as onset of confirmed objective response as per Investigator assessment according to the RECIST 1.0 criteria.
Time Frame: Response determined during Stage 2 or within 28 days after termination of Stage 2 treatment
Population: Patients treated in Stage 2
Measure: Number; unit: Number of participants
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 1 | 2
Number of participants
  Week 2 (Day 1 - 14) | 0 | 0
  Week 4 (Day 15 - 56) | 1 | 1
  Week 12 (Day 57 - 112) | 0 | 1

10. Secondary Outcome: Best RECIST Assessment as Confirmed Duration of Objective Response and Disease Control as Per Investigator Assessment for Stage 1
Description: Best RECIST Assessment as duration of confirmed objective response and disease control as per Investigator assessment according to the RECIST 1.0 criteria.
Time Frame: as for outcome 3
Population: Randomised Set (RS)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
Weeks
  Duration of objective response (N=10; N=4) | 21.4 (12.2) | 58.9 (98.1)
  Duration of disease control(N=31; N=35) | 25.1 (13.9) | 30.3 (35.8)

11. Secondary Outcome: Best RECIST Assessment as Confirmed Duration of Confirmed Objective Response and Disease Control as Per ICR for Stage 1
Description: Best RECIST Assessment as duration of confirmed objective response and disease control as per the independent central review (ICR) according to the RECIST 1.0 criteria.
Time Frame: as for outcome 3
Population: Randomised Set (RS)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
Weeks
  Duration of objective response (N=5; N=6) | 28.0 (12.6) | 55.1 (76.6)
  Duration of disease control(N=29; N=30) | 22.8 (11.0) | 28.8 (38.1)

12. Secondary Outcome: Best RECIST Assessment as Confirmed Duration of Objective Response and Disease Control as Per Investigator Assessment for Stage 2
Description: Best RECIST Assessment as confirmed duration of objective response and disease control as per Investigator assessment according to the RECIST 1.0 criteria.
Time Frame: Response determined during Stage 2 or within 28 days after termination of Stage 2 treatment
Population: patients treated in stage 2
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 36 | 32
Weeks
  Duration of objective response (N=1; N=2) | 24.7 (0.0) | 19.4 (21.1)
  Duration of disease control(N=14; N=6) | 21.8 (6.1) | 21.5 (12.3)

13. Secondary Outcome: Best RECIST Assessment as Confirmed Duration of Disease Control as Per ICR for Stage 2
Description: Best RECIST Assessment as confirmed duration of disease control as per the independent central review (ICR) assessment according to the RECIST 1.0 criteria.
Time Frame: Response determined during Stage 2 or within 28 days after termination of Stage 2 treatment
Population: patients treated in stage 2
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab 250 mg/m2 - Stage 2
Number analyzed (Participants) | 36 | 32
Weeks | 17.4 (5.0) | 18.4 (10.0)

14. Secondary Outcome: Progression Free Survival (PFS) Before Crossover Based on Investigator Assessment
Description: PFS is defined as time from randomisation to until the occurrence of tumor progression or death, whichever occurred first, during Stage 1 of the trial.
  Median is calculated from the Kaplan-Meier curve for each treatment group.
Time Frame: From randomisation to disease progression in Stage 1 or death whichever occurred first before crossover.
Population: Randomised set (RS).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab 250 mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
weeks | 15.86 [10.29 to 17.14] | 15.14 [8.29 to 19.29]
Statistical Analysis 1: Comparison: Afatinib 50 mg - Stage 1 vs Cetuximab 250 mg/m2 - Stage 1; Test type: Superiority or Other; p = 0.764, Regression, Cox; Hazard Ratio (HR) = 0.942, 95% CI 2-sided [0.640 to 1.387] — Hazard ratio, 95% CI and p-value are calculated from the Cox proportional hazards model stratified by the number of prior chemotherapies for R/M setting (0 or >=1)

15. Secondary Outcome: Progression Free Survival (PFS) After Crossover Based on Investigator Assessment
Description: PFS is defined as time from first administration study medication after cross over until the occurrence of tumor progression or death, whichever came first, during Stage 2 of the trial.
  Median is calculated from the Kaplan-Meier curve for each treatment group.
Time Frame: From first administration of study medication after cross over to disease progression in Stage 2 or death whichever came first after crossover.
Population: Patients treated in stage 2
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Cetuximab mg/m2 - Stage 2: Patients were randomized to Afatinib monotherapy 50mg once daily (q.d.) in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week (load) followed by 250mg/m2 weekly thereafter in Stage 2.
Arm/Group | Afatinib 50 mg - Stage 2 | Cetuximab mg/m2 - Stage 2
Number analyzed (Participants) | 36 | 32
weeks | 7.93 [4.29 to 14.43] | 6.43 [4.14 to 8.29]
Statistical Analysis 1: Comparison: Afatinib 50 mg - Stage 2 vs Cetuximab mg/m2 - Stage 2; Test type: Superiority or Other; p = 0.219, Regression, Cox; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.434 to 1.212] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomisation to death.
  Median is calculated from the Kaplan-Meier curve for each treatment group.
Time Frame: From randomisation to data cut-off date.
Population: Randomised set (RS).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Afatinib 50 mg / Cetuximab 250mg/m2 | Cetuximab 250 mg/m2 / Afatinib 50 mg
Number analyzed (Participants) | 62 | 62
Weeks | 35.86 [25.71 to 45.00] | 47.14 [24.14 to 64.71]
Statistical Analysis 1: Comparison: Afatinib 50 mg / Cetuximab 250mg/m2 vs Cetuximab 250 mg/m2 / Afatinib 50 mg; Test type: Superiority or Other; p = 0.758, Regression, Cox; Hazard Ratio (HR) = 1.067, 95% CI 2-sided [0.708 to 1.608] — [estimate comment as in outcome 14, analysis 1]

17. Secondary Outcome: Time to Deterioration in HRQoL - Stage 1
Description: Health related Quality of Life (HRQoL) for Time to deterioration was assessed using the the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the Head and Neck Cancer Module (H&N35).
  Time to deterioration in HRQoL (defined as a 10-point change towards worsening from the baseline score on a 0-100 point scale) was determined for:
  * global health status (Questions 29 and 30 in EORTC QLQ C30)
  * pain (Questions 9 and 19 in EORTC QLQ C30)
  * swallowing (Questions 35 to 38 in EORTC QLQ-H&N35)
Time Frame: From randomisation to deterioration in HRQoL scores before crossover.
Population: Randomised Set (RS)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Afatinib 50 mg - Stage 1: Patients were randomised to receive Afatinib 50 mg in stage 1
- Cetuximab mg/m2 - Stage 1: Patients were randomized to Cetuximab 250 mg/m2 received 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab mg/m2 - Stage 1
Number analyzed (Participants) | 62 | 62
months
  global health status (N=37; N=38) | 2.83 [1.91 to 5.85] | 3.94 [2.96 to 7.39]
  pain (N=34; N=33) | 2.73 [1.48 to 5.88] | 4.63 [2.92 to 8.61]
  swallowing (N=33; N=34) | 5.59 [2.07 to 7.36] | 6.60 [2.92 to 8.48]

18. Secondary Outcome: Patients With AEs Resulting in Diarrhea, Skin Rash, Dose Reduction, Treatment Discontinuation and Decreased Cardiac Left Ventricular Function
Description: Patients with adverse events (AEs) resulting in Diarrhea, Skin Rash, dose reduction, treatment discontinuation and decreased cardiac left ventricular function
  Note: To asses the Decreased Cardiac left ventricular function, Left ventricular ejection fraction (LVEF) was assessed in patients treated with afatinib in Stage 1 and Stage 2 . And no patients in either group had a significant change in LVEF during Stage 1 or Stage 2 of the trial.
Time Frame: First administration of trial medication until 28 days after last drug administration
Population: Treated Set in Stage 1 : This analysis set included the randomized patients who took at least 1 dose of the randomized treatment (61 afatinib and 60 cetuximab patients. Treated set in Stage 2: This analysis set included all patients who received treatment: 36 patients in the afatinib and 32 patients in the cetuximab arm.
Measure: Number; unit: number of participants
Groups:
- Afatinib 50 mg - Stage 2: Patients were randomized to Cetuximab 250 mg/m2 received 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Afatinib 50 mg once daily (q.d.) for Stage 2
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab mg/m2 - Stage 1 | Afatinib 50 mg - Stage 2 | Cetuximab mg/m2 - Stage 2
Number analyzed (Participants) | 61 | 60 | 36 | 32
number of participants
  With AE leading to Diarrhea | 49 | 15 | 22 | 2
  With AE leading to skin rash | 48 | 46 | 23 | 14
  With AE leading to dose reduction | 18 | 2 | 11 | 0
  With AE leading to treatment discontinuation | 23 | 11 | 8 | 6

19. Secondary Outcome: Incidence and Intensity of Adverse Events With Grading According CTCAE
Description: Incidence and intensity of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: First administration of trial medication until 28 days after last drug administration
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 50 mg - Stage 1 | Cetuximab mg/m2 - Stage 1 | Afatinib 50 mg - Stage 2 | Cetuximab mg/m2 - Stage 2
Number analyzed (Participants) | 61 | 60 | 36 | 32
percentage of participants
  CTCAE grade 1 | 3.3 | 5.0 | 5.6 | 9.4
  CTCAE grade 2 | 24.6 | 41.7 | 25.0 | 37.5
  CTCAE grade 3 | 39.3 | 28.3 | 25.0 | 25.0
  CTCAE grade 4 | 8.2 | 6.7 | 13.9 | 9.4
  CTCAE grade 5 | 24.6 | 16.7 | 30.6 | 15.6

20. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma for Dose 40mg and 50mg at Steady State on Day 15 (Cpre,ss,15)
Description: Cpre,ss,15 represents the pre-dose concentration of afatinib in plasma at steady state on day 15.
  Note: At day 15, values for afatinib 40 mg no values reported in stage 1 and stage 2.
Time Frame: Day 15
Population: Pharmacokinetic Set (PK): The PK analysis was based on all patients who were treated with afatinib and who had evaluable plasma concentration data, which consisted of data for 60 patients in Stage 1 and 35 patients in Stage 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 50 mg - Stage 1 | Afatinib 50 mg - Stage 2
Number analyzed (Participants) | 45 | 26
ng/mL | 39.3 (70.1) | 46.6 (81.4)

21. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma for Dose 40mg and 50mg at Steady State on Day 29 (Cpre,ss,29)
Description: Cpre,ss,29 represents the pre-dose concentration of afatinib in plasma at steady state on day 29.
  Note: At day 29, values for afatinib 40 mg no values reported in stage 2.
Time Frame: Day 29
Population: Pharmacokinetic Set (PK)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 40 mg - Stage 1: Patients were randomised to receive Afatinib 50 mg once daily (q.d.) in Stage 1, and had sequential dose reduction to 40 mg in stage 1.
Arm/Group | Afatinib 40 mg - Stage 1 | Afatinib 50 mg - Stage 1 | Afatinib 50 mg - Stage 2
Number analyzed (Participants) | 9 | 33 | 22
ng/mL | 8.84 (206) | 31.7 (97.7) | 45.9 (48.9)

22. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma for Dose 40mg and 50mg at Steady State on Day 57 (Cpre,ss, 57)
Description: Cpre,ss,57 represents the pre-dose concentration of afatinib in plasma at steady state on day 57.
Time Frame: Day 57
Population: Pharmacokinetic Set (PK)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 40 mg - Stage 1 | Afatinib 50 mg - Stage 1 | Afatinib 50 mg - Stage 2
Number analyzed (Participants) | 7 | 16 | 10
ng/mL | 32.7 (25.3) | 19.9 (94.4) | 46.5 (67.2)

ADVERSE EVENTS:
Time Frame: 1493 days
Groups:
- Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 1; Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 2: Patients were randomized to Cetuximab 250 mg/m2 received 400mg/m2 once in the first week followed by 250 mg/m2 weekly thereafter in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Afatinib 50 mg once daily (q.d.) for Stage 2.
- Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 2; Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 1: Patients were randomized to Afatinib monotherapy 50mg once daily (q.d.) in Stage 1 and if the patients had disease progression or intolerable AEs were crossed over to Cetuximab 250 mg/m2 given as 400mg/m2 once in the first week (load) followed by 250mg/m2 weekly thereafter in Stage 2.
Arm/Group | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 1 | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 2 | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 2 | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 1
Serious Adverse Events (participants affected / at risk) | 26/60 | 18/36 | 13/32 | 36/61
Other Adverse Events (participants affected / at risk) | 59/60 | 34/36 | 29/32 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 1 (N=60) | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 2 (N=36) | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 2 (N=32) | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 1 (N=61)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 2
Endocarditis noninfective (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 8
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 2
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 3 | 6 | 3 | 6
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 2 | 0
Meningitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 5
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 8
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Linitis plastica (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 3
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 3
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 1 (N=60) | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 2 (N=36) | Cetuximab 250 mg/m2 / Afatinib 50 mg - Stage 2 (N=32) | Afatinib 50 mg / Cetuximab 250mg/m2 - Stage 1 (N=61)
Anaemia (Blood and lymphatic system disorders) | 10 | 3 | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 7 | 4 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 4
Cheilitis (Gastrointestinal disorders) | 2 | 1 | 0 | 4
Constipation (Gastrointestinal disorders) | 17 | 2 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 15 | 21 | 2 | 45
Dry mouth (Gastrointestinal disorders) | 5 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 2 | 1 | 6
Nausea (Gastrointestinal disorders) | 17 | 8 | 2 | 22
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 4 | 0 | 5
Vomiting (Gastrointestinal disorders) | 12 | 7 | 1 | 15
Asthenia (General disorders) | 9 | 3 | 4 | 10
Fatigue (General disorders) | 19 | 5 | 6 | 18
Mucosal inflammation (General disorders) | 11 | 7 | 1 | 14
Pyrexia (General disorders) | 11 | 3 | 3 | 4
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 4
Paronychia (Infections and infestations) | 4 | 3 | 2 | 3
Upper respiratory tract infectio (Infections and infestations) | 1 | 2 | 1 | 1
Weight decreased (Investigations) | 8 | 5 | 1 | 9
Decreased appetite (Metabolism and nutrition disorders) | 11 | 7 | 6 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1 | 0 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 3
Dizziness (Nervous system disorders) | 7 | 1 | 1 | 5
Headache (Nervous system disorders) | 5 | 3 | 5 | 4
Paraesthesia (Nervous system disorders) | 1 | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 2
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 4
Insomnia (Psychiatric disorders) | 5 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 3 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 8 | 3 | 4 | 8
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 3 | 3 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 4 | 3 | 9
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 8
Rash (Skin and subcutaneous tissue disorders) | 25 | 10 | 6 | 26
Skin fissures (Skin and subcutaneous tissue disorders) | 11 | 1 | 1 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 2
Xeroderma (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 4
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication